CLINICAL TRIAL: NCT04813653
Title: A Single-arm, Prospective Study of Cyclosporine in Combination With Carfilzomib and Dexamethasone in Patients With Relapsed Multiple Myeloma Refractory to Carfilzomib With High Expression of the Peptidylprolyl Isomerase A (PPIA) Gene in Myeloma Cells
Brief Title: Cyclosporine in Combination With Carfilzomib and Dexamethasone in Relapsed Multiple Myeloma Refractory to Carfilzomib and High Expression of PPIA Gene in Myeloma Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1007-20-TLV
Record Dates: First submitted 2021-03-18; First posted 2021-03-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclosporine; carfilzomib; Dexamethasone

STUDY DESIGN:
Intervention Model Description: single-arm, prospective study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cyclosporine in combination with carfilzomib and dexamethasone (Experimental): cyclosporine in combination with carfilzomib and dexamethasone in patients with relapsed multiple myeloma refractory to carfilzomib with high expression of the PPIA gene in myeloma cells
  Interventions: Drug: cyclosporine in combination with carfilzomib and dexamethasone

INTERVENTIONS:
Drug: cyclosporine in combination with carfilzomib and dexamethasone — patients will be treated with cyclosporine with dose titration based on repeated determinations of whole blood concentrations to achieve a target trough concentration of 250 ng/mL, in combination with carfilzomib plus dexamethasone.

SUMMARY:
This phase 1, open-label, single-arm, prospective, single center study will evaluate the safety, tolerability and efficacy of cyclosporine in combination with carfilzomib and dexamethasone in patients with relapsed and refractory multiple myeloma (RRMM).

DETAILED DESCRIPTION:
This phase 1, open-label, single-arm, prospective, single center study will evaluate the safety, tolerability and efficacy of cyclosporine in combination with carfilzomib and dexamethasone in patients with relapsed and refractory multiple myeloma (RRMM). The patients will consist of adult men and women who have a confirmed diagnosis of RRMM, who have received at least two prior lines of therapy including carfilzomib, and were non responsive or refractory to carfilzomib as specified below, and who were found to have elevated expression of Peptidylprolyl Isomerase A (PPIA) in scRNA sequencing of their myeloma cells, and who meet other protocol outlined eligibility criteria.

The patients will be treated with cyclosporine with dose titration based on repeated determinations of whole blood concentrations to achieve a target trough concentration of 250 ng/mL, in combination with carfilzomib plus dexamethasone.

Patients may continue to receive treatment for 4 months or until disease progression or unacceptable toxicity, the earliest of them.

Subjects will be followed for Adverse Events (AEs), clinical status-Overall response rate (ORR) as defined by International Myeloma Working Group (IMWG) criteria, Progression Free Survival (PFS), Duration of Response (DOR), Time to Progression (TTP), stringent Complete Response (sCR 0, Complete Response (CR), Very Goog Partial Response (VGPR), Partial Response (PR), Depth of Best Response (DpR), Time To Response (TTR), Progressive Disease (PD), Overall Survival (OS) and laboratory parameters for up to 4 months, unless they terminate early due to disease progression, unacceptable toxicity or due to meeting one of the withdrawal criteria

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria:

1. Male or female patients, 18 years of age or older.
2. Multiple myeloma diagnosed according to standard IMWG criteria.
3. Patients must have measurable disease defined by at least one of the following three measurements:

   * Serum M-protein 1 g/dL (10 g/L).
   * Urine M-protein 200 mg/24 hours.
   * Serum free light chain assay: involved free light chain level at least 100 mg/L, provided that the serum free light chain ratio is abnormal.
4. Patients received one or two prior lines of therapy which must have included bortezomib, lenalidomide-and daratumumab.
5. Patient received carfilzomib-based therapy either as their most recent line of therapy and within 3 months from study enrolment, and either failed to achieve a minor response after completing 2 cycles of carfilzomib based therapy, or are refractory to treatment.
6. Patients were found to have a high-expression level of PPIA, >1.2 unique RNA molecules (UMI) per cell on average, by scRNA sequencing of their myeloma cells from bone marrow aspiration sample at study screening.
7. Patients must meet the following clinical laboratory criteria:

   * Absolute neutrophil count (ANC) ≥1,000/mm3 and platelet count≥75,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days of enrolment.
   * Total bilirubin ≤1.5 the upper limit of the normal range (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 ULN.
   * Calculated creatinine clearance ≥45 mL/min
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
9. Female patients who:

   * Are postmenopausal for at least 24 months before the screening visit, OR
   * Are surgically sterile, OR
   * Who are of childbearing potential, and agree to practice two effective methods of contraception (1 highly effective method and 1 additional effective method) at the same time, from the time of signing the informed consent through 90 days after the last dose of study treatment, OR agree to completely abstain from heterosexual intercourse.

   Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 milli International Units/mL within 10 to 14 days of initiation of Cycle 1 and again within 24 hours of starting Cycle 1. FCBP must also agree to ongoing pregnancy testing. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
10. Male patients, even if surgically sterilized (i.e., status postvasectomy), who:

    * Agree to completely abstain from heterosexual intercourse, OR
    * Agree to practice effective barrier contraception (i.e., latex condom) during sexual contact with a FCBP, even if they have had a successful vasectomy, throughout the entire study treatment period and through 4 months after the last dose of study treatment.
11. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
12. Patient is willing and able to adhere to the study visit schedule and other protocol requirements.

    -

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria are not eligible to participate in the study:

  1. Patient underwent an allogeneic transplantation.
  2. Major surgery within 14 days before enrolment.
  3. Central nervous system involvement
  4. Concomitant use of any other antineoplastic treatment with activity against MM (with the exception of ≤40 mg Dexamethasone per day or equivalent for no longer than 4 days).
  5. Anti-myeloma therapy as follows prior to screening bone marrow aspiration:

     1. Targeted therapy, within 14 days or at least 5 half-lives, whichever is less;
     2. Monoclonal antibody treatment for multiple myeloma within 21 days;
     3. Cytotoxic therapy within 14 days;
     4. Proteasome inhibitor therapy within 14 days; note: no window is required for carfilzomib
     5. Immunomodulatory agent therapy within 7 days.
     6. Radiotherapy within 14 days (with the exception of radiotherapy for spinal cord compression or for pain control that should be discussed and approved by the sponsor- investigator prior to study enrolment). However, if the radiation portal covered ≤5% of the bone marrow reserve, the subject is eligible irrespective of the end date of radiotherapy.
  6. Diagnosed or treated for another malignancy within 2 years before enrolment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
  7. Moderate to severe kidney injury (Calculated creatinine clearance ≤45 mL/min).
  8. Severe liver disease (cirrhosis grade Child-Pugh B or C; significant hepatocellular or cholestatic liver injury).
  9. Diagnosis of Waldenstrom's macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes) syndrome, plasma cell leukaemia, primary amyloidosis, myelodysplastic syndrome, or myeloproliferative syndrome.
  10. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
  11. Psychiatric illness/social situation that would limit compliance with study requirements.
  12. Patient with a known diagnosis of Epilepsy.
  13. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
  14. Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
  15. Systemic treatment with strong inhibitors of Cytochrome P450 family 3, subfamily A (CYP3A) (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong Cytochrome P450 (CYP3A), family 3, subfamily A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort within 14 days before enrolment in the study.
  16. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before enrolment.
  17. Ongoing or active systemic infection, active hepatitis B virus infection, active hepatitis C infection, or known human immunodeficiency virus (HIV) positive.
  18. Vaccination with live attenuated viruses (i.e. yellow fever injections, polio drops, chickenpox (herpes varicella) and shingles (herpes zoster) vaccines) within 30 days before enrolment.
  19. Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or known GI disease or planned gastrointestinal (GI) procedure that could interfere with the oral absorption or tolerance of treatment.
  20. Failure to have fully recovered (ie, Grade 1 toxicity) from the reversible effects of prior chemotherapy (except for alopecia).
  21. Patient has Grade 3 peripheral neuropathy during the screening period.
  22. Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.
  23. Patients that have previously been treated with Cyclosporine plus carfilzomib.
  24. Female patients who are lactating or pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-04-18 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment parameters. | follow-up 2 years post study
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment parameters.

SECONDARY OUTCOMES:
Overall response rate ORR | follow-up 2 years post study
  Proportion of patients who achieve a best overall response of stringent complete response , complete response, very good partial response, or partial response as defined using the IMWG criteria
Progression free survival PFS | follow-up 2 years post study
  The time from first dose to the date of the first documented tumor progression or death due to any cause. PFS will be determined by an investigator, based upon laboratory data, as defined by the IMWG criteria
Duration of Response DOR | follow-up 2 years post study
  The time between the date of first response to the date of the first objectively documented tumor progression as assessed by study steering committee according to modified IMWG criteria or death due to any cause prior to subsequent anti-cancer therapy.
Time to Response TTR | follow-up 2 years post study
  The time from the first dose to the date of the first sCR, CR, VGPR, or PR.
Depth of Best Response (DpR) | follow-up 2 years post study
  According to IMWG criteria.
Time to progression (TTP) | follow-up 2 years post study
  Time from initiation of treatment to documented PD
Overall Survival (OS) | follow-up 2 years post study
  Time between the date of first dose and the date of death due to any cause
Extramedullary progression | follow-up 2 years post study
  Kaplan Meyer test will be applied to test for differences between the groups in Progression Free Survival
Extramedullary progression | follow-up 2 years post study
  Kaplan Meyer test will be applied to test for differences between the groups in Overall Survival
Percentage of cyclosporine trough levels tests in acceptable range | follow-up 2 years post study
  will be calculated for each patient.
Mean % of levels in acceptable range will be calculated for the efficacy population. | follow-up 2 years post study

CONTACTS AND LOCATIONS:
Overall Officials: Yael Cohen, MD, Principal Investigator — TASMC
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No